CLINICAL TRIAL: NCT05915741
Title: Brain Recordings in Patients Undergoing Deep Brain Stimulation (DBS) for Severe Obsessive-Compulsive Disorder (OCD)
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sameer Sheth, Professor, Baylor College of Medicine
Other Study IDs: H-48392
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Obsessive-compulsive disorder effects approximately 2-3% of the population. The only established first-line treatments for OCD are cognitive-behavioral therapy (CBT) with exposure/response prevention and serotonin reuptake inhibitor medications (SRIs). Approximately 30-40% of patients fail to respond to either modality and few patients experience complete symptom resolution. Up to 25% of patients have difficulty tolerating CBT, and the risk of relapse after therapies remains significant. Symptoms of OCD include unwanted, distressing thoughts and rituals such as excessive washing of hands or other body parts, rechecking things such as locks or switches because of obsessional doubt, and avoidance of anxiety-provoking situations. In some cases, compulsions can consume several hours per day and in the most extreme cases can involve most of the patient's waking hours (e.g. washing hands hundreds of times per day, 18-hour showers). Medical complications may result from repeated washing or other repetitive behaviors. Significant social and occupational impairment can result from this disorder and some patients are housebound or even bed-ridden.

Effective evidence-based treatments include behavior therapy and certain medications. Despite these therapies, a significant number of patients are treatment resistant and suffer persistent, debilitating symptoms. In severe cases, neurosurgical intervention is sometimes performed to alleviate symptoms. A common surgical option is deep brain stimulation (DBS), a procedure that involves placing two electrodes in a specific region in the brain and connecting them to a pacemaker-like device implanted under the skin in the upper chest. The clinician adjusts the stimulation parameters on the device to find the settings that best relieve symptoms.

One of the challenges of treating a psychiatric disorder is the absence of reliable and valid biomarkers for diagnosing and objectively monitoring treatment outcomes. There is also problem of heterogeneity, which introduces additional barriers to predicting who will respond best to a particular treatment. A better understanding of the dysfunction in key brain circuits underlying OCD symptomatology will allow us to improve outcomes with DBS. The pathophysiology of OCD is associated with dysfunction in prefrontal cortico-basal ganglia circuits. The electrodes of the DBS system are placed at a critical hub within this circuit. This target is called the ventral capsule/ventral striatum (VC/VS). DBS targeting the VC/VS is approved for the treatment of severe OCD under an FDA Humanitarian Device Exemption (HDE).

In this project, the investigators will recruit patients treated with DBS for OCD under the standard clinical (HDE) pathway. The FDA/HDE-approved device for these procedures is the Medtronic Percept DBS system. The Percept implanted pulse generator (IPG; pacemaker-like device mentioned above that delivers stimulation) has the ability to not only stimulate, but also record electrical activity measured from the brain electrodes, store the recordings in memory, and wirelessly transmit them to the clinician. The investigators will ask consenting patients to perform and transmit these recordings to the investigators for analysis. The investigators hope that these recordings will help them understand the relationship between electrical network activity in the brain and patient symptoms. A closer understanding of this relationship may eventually enable the investigators to make better informed programming adjustments and therefore achieve better symptom control.

The main objective is to obtain recordings from the VC/VS, a key network hub in OCD, in patients already implanted with a DBS system for severe OCD. The Investigators will use these recordings to better understand the relationship between brain activity and OCD symptoms, with the hope that this understanding will lead to more effective utilization of DBS therapy to treat severe OCD.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years old or older
* Implanted with the Medtronic Percept DBS system to treat OCD

Exclusion Criteria:

* Unable to operate the patient programmer to perform recordings
* Unable to provide informed consent

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Subjects whom are implanted with the Medtronic Percept DBS system for OCD will be enrolled.
Sampling Method: Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Y-BOCS (Yale-Brown Obsessive Compulsive Scale) score | 12 months
  0: <25% reduction in Y-BOCS scores (non-response), 1: 25-35% Y-BOCS score reduction (partial response), 2: ≥35% Y-BOCS score reduction (response), 3: ≥35% Y-BOCS score reduction and final Y-BOCS ≤ 12 (remitter).
  Lower scores equal better outcome. Minimum value: 0 Maximum value: 50

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No